CLINICAL TRIAL: NCT04493281
Title: Bioequivalence Study of Oral Suspension and Intravenous Formulation of Edaravone in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MT-1186-J03
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Edaravone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT-1186 (Experimental): Healthy subjects were administered a single dose of Edaravone oral suspension
  Interventions: Drug: MT-1186
- MCI-186 (Active Comparator): Healthy subjects were administered a single dose of Edaravone intravenous formulation
  Interventions: Drug: MCI-186

INTERVENTIONS:
Drug: MT-1186 — Oral suspension
  Other Names: Edaravone
  Arms: MT-1186
Drug: MCI-186 — Intravenous formulation
  Other Names: Edaravone
  Arms: MCI-186

SUMMARY:
To evaluate the single-dose bioequivalence of oral suspension and intravenous (IV) formulation of edaravone in the fasting state in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteers
* Japanese
* Subjects aged between 20 and 45 years at the time of informed consent
* Subjects who have thoroughly understood the contents of the study and voluntarily provided written informed consent to participate in the study

Exclusion Criteria: Additional screening criteria check may apply for qualification:

* Subjects with a current or previous history of cardiac, hepatic, renal, gastrointestinal, respiratory, psychiatric/nervous, hematopoietic, or endocrine diseases, and those whom the investigator (or subinvestigator) deems unsuitable for the study
* Body mass index (BMI) of <18.0 or >30.0, or body weight of <50 kg (BMI formula: body weight [kg]/height [m]2, rounded to one decimal place)
* Subjects who have undergone any surgery known to affect the gastrointestinal absorption of drugs
* Female subjects who do not agree to use an effective method of contraception from screening or 2 weeks before the start of investigational product administration, whichever comes earlier, to 14 days after the completion (or discontinuation) of investigational product administration. Male subjects who do not agree to use an effective method of contraception from the start of investigational product administration to 14 days after the completion (or discontinuation) of investigational product administration
* Subjects who have previously received edaravone
* Subjects who have participated in another clinical study and received an investigational product within 12 weeks before providing informed consent

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-04-21 (Actual); Study Completion 2019-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shimizu H, Nishimura Y, Shiide Y, Yoshida K, Hirai M, Matsuda M, Nakamaru Y, Kato Y, Kondo K. Bioequivalence Study of Oral Suspension and Intravenous Formulation of Edaravone in Healthy Adult Subjects. Clin Pharmacol Drug Dev. 2021 Oct;10(10):1188-1197. doi: 10.1002/cpdd.952. Epub 2021 May 6. PMID 33955162

RESULTS

PARTICIPANT FLOW:
Groups:
- Edaravone Oral Suspensione First, Then Edaravone IV Formulation: Period 1: a single dose of Edaravone oral suspension (105 mg) . Period 2: a single dose of Edaravone IV formulation (60 mg/60 min).
- Edaravone IV Formulation First, Then Edaravone Oral Suspension: Period 1: a single dose of Edaravone IV formulation (60 mg/60 min). Period 2: a single dose of Edaravone oral suspension (105 mg) .
Period: Period 1
Arm/Group | Edaravone Oral Suspensione First, Then Edaravone IV Formulation | Edaravone IV Formulation First, Then Edaravone Oral Suspension
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Edaravone Oral Suspensione First, Then Edaravone IV Formulation | Edaravone IV Formulation First, Then Edaravone Oral Suspension
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edaravone Oral Suspensione First, Then Edaravone IV Formulation | Edaravone IV Formulation First, Then Edaravone Oral Suspension | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 21 | 21 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero up to the Last Quantifiable Concentration Time-point (AUC0-t) of Unchanged Edaravone After Oral and Intravenous Administration
Time Frame: The date of dosing is defined as Day 1. PO: Day 1 at pre-dose, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12 hrs; IV: Day 1 at pre-dose, 0.25, 0.5, 1, 1.083, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12 hrs; Both groups: Day 2 at 24, 36 hrs; Day 3 at 48 hrs.
Population: This study was designed as a 2-group, 2-period crossover study with the advance administration of edaravone oral suspension group (PO => IV) with 21 subjects, and the advance administration of edaravone IV formulation group (IV => PO) with 21 subjects to investigate the bioequivalence between edaravone oral suspension and edaravone IV formulation.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Groups:
- Edaravone Oral Suspension: Healthy subjects were administered a single dose of Edaravone oral suspension (105 mg) under fasted condition.
- Edaravone IV Formulation: Healthy subjects were administered a single dose of Edaravone IV formulation (60 mg/60 min) under fasted condition.
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
ng·h/mL | 1743 (534) | 1720 (326)
Statistical Analysis 1: Comparison: Edaravone Oral Suspension vs Edaravone IV Formulation; Test type: Equivalence — The analysis was performed by analysis of variance (ANOVA), which included factors accounting for the following sources of variation: sequence, subjects nested in sequences, period, and treatment. For bioequivalence, the 90% CIs of the geometric mean ratio of AUC0-t for oral suspension and intravenous formulation were required to be within the range of 0.80 to 1.25; Ratio (PO/IV) = 0.97, 90% CI 2-sided [0.91 to 1.04]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero up to Infinity With Extrapolation of the Terminal Phase (AUC0-inf) of Unchanged Edaravone After Oral and Intravenous Administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
ng·h/mL | 1762 (540) | 1736 (331)
Statistical Analysis 1: Comparison: Edaravone Oral Suspension vs Edaravone IV Formulation; Test type: Equivalence — The analysis was performed by analysis of variance (ANOVA), which included factors accounting for the following sources of variation: sequence, subjects nested in sequences, period, and treatment. For bioequivalence, the 90% CIs of the geometric mean ratio of AUC0-inf for oral suspension and intravenous formulation were required to be within the range of 0.80 to 1.25; Ratio (PO/IV) = 0.98, 90% CI 2-sided [0.92 to 1.04]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Unchanged Edaravone After Oral and Intravenous Administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
ng/mL | 1656 (733.6) | 1253 (228.9)
Statistical Analysis 1: Comparison: Edaravone Oral Suspension vs Edaravone IV Formulation; Test type: Equivalence — The analysis was performed by analysis of variance (ANOVA), which included factors accounting for the following sources of variation: sequence, subjects nested in sequences, period, and treatment. For bioequivalence, the 90% CIs of the geometric mean ratio of Cmax for oral suspension and intravenous formulation were required to be within the range of 0.80 to 1.25; Ratio (PO/IV) = 1.22, 90% CI 2-sided [1.09 to 1.36]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
h
  Unchanged edaravone | 0.50 [0.25 to 0.75] | 1.00 [0.98 to 1.02]
  Sulfate conjugate | 0.75 [0.50 to 1.00] | 1.08 [0.98 to 1.25]
  Glucuronide Conjugate | 0.75 [0.25 to 1.00] | 1.08 [1.00 to 1.27]

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero up to 24 Hours (AUC0-24)
Time Frame: The date of dosing is defined as Day 1. PO: Day 1 at pre-dose, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12 hrs; Day 2 at 24 hrs ; IV: Day 1 at pre-dose, 0.25, 0.5, 1, 1.083, 1.25, 1.5, 1.75,2, 3, 4, 6, 8, 12 hrs; Day 2 at 24 hrs.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
ng·h/mL
  Unchanged edaravone | 1735 (523) | 1714 (317)
  Sulfate conjugate | 19837 (5185) | 14830 (3519)
  Glucuronide Conjugate | 3917 (727) | 2288 (479)

6. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero up to the Last Sampling Time-point (for All Time-points) (AUC0-all)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
ng·h/mL
  Unchanged edaravone | 1752 (532) | 1727 (323)
  Sulfate conjugate | 20035 (5252) | 15025 (3575)
  Glucuronide Conjugate | 3927 (730) | 2297 (481)

7. Secondary Outcome: Terminal Elimination Half-life (t1/2)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
h
  Unchanged edaravone | 9.75 (8.47) | 8.82 (8.33)
  Sulfate conjugate | 5.77 (1.85) | 7.58 (2.39)
  Glucuronide Conjugate | 3.75 (0.55) | 3.69 (0.48)

8. Secondary Outcome: Elimination Rate Constant From the Central Compartment (Kel)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
1/h
  Unchanged edaravone | 0.1194 (0.0876) | 0.1156 (0.0563)
  Sulfate conjugate | 0.1295 (0.0318) | 0.1010 (0.0324)
  Glucuronide Conjugate | 0.1909 (0.0417) | 0.1924 (0.038)

9. Secondary Outcome: Mean Residence Time From Time Zero up to Infinity With Extrapolation of the Terminal Phase (MRT0-inf) of Unchanged Edaravone
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
h | 2.495 (0.903) | 2.333 (0.826)

10. Secondary Outcome: Total Clearance (CL) of Unchanged Edaravone After Intravenous Administration
Time Frame: The date of dosing is defined as Day 1. Day 1 at pre-dose, 0.25, 0.5, 1, 1.083, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12 hrs; Day 2 at 24, 36 hrs; Day 3 at 48 hrs.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Edaravone IV Formulation
Number analyzed (Participants) | 42
L/h | 35.9 (7.5)

11. Secondary Outcome: Volume of Distribution During Terminal Phase (Vz) of Unchanged Edaravone After Intravenous Administration
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Edaravone IV Formulation
Number analyzed (Participants) | 42
L | 418 (321)

12. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Unchanged Edaravone After Intravenous Administration
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Edaravone IV Formulation
Number analyzed (Participants) | 42
L | 63.1 (22.0)

13. Secondary Outcome: Apparent Total Clearance (CL/F) of Unchanged Edaravone After Oral Administration
Time Frame: The date of dosing is defined as Day 1. Day 1 at pre-dose, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12 hrs; Day 2 at 24, 36 hrs; Day 3 at 48 hrs.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Edaravone IV Formulation
Number analyzed (Participants) | 42
L/h | 67.9 (30.1)

14. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) of Unchanged Edaravone After Oral Administration
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Edaravone Oral Suspension
Number analyzed (Participants) | 42
L | 826 (618)

15. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss/F) of Unchanged Edaravone After Oral Administration
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Edaravone Oral Suspension
Number analyzed (Participants) | 42
L | 164.0 (78.9)

16. Secondary Outcome: Cumulative Amount of Drug Excreted in Urine From Time Zero up to 48 Hours (Ae0-48)
Time Frame: Urine samples are collected: Day1 to 6.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
mg
  Unchanged edaravone | 0.66 (0.21) | 0.52 (0.15)
  Sulfate conjugate | 10.04 (8.67) | 7.06 (6.43)
  Glucuronide Conjugate | 125.9 (19.0) | 94.3 (13.7)

17. Secondary Outcome: Cumulative Percentage of Drug Excreted in Urine From Time Zero up to 48 Hours (Ae0-48)
Time Frame: Urine samples are collected: Day1 to 6.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
percentage of dose
  Unchanged edaravone | 0.629 (0.199) | 0.869 (0.252)
  Sulfate conjugate | 6.58 (5.68) | 8.09 (7.37)
  Glucuronide Conjugate | 59.8 (9.0) | 78.4 (11.4)

18. Secondary Outcome: Renal Clearance (CLr) of Unchanged Edaravone
Time Frame: Urine samples are collected: Day1 to 6.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
L/h | 0.424 (0.227) | 0.311 (0.114)

19. Secondary Outcome: Bioavailability (F) of Unchanged Edaravone After Oral Administration
Description: Bioavailability was calculated from ratio of AUC0-inf of unchanged edaravone after oral and intravenous administration.
Time Frame: PO: Day 1 at pre-dose, 0.083, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, and 12 hrs; Day 2 at 24 and 36 hrs; Day 3 at 48 hrs. IV: Day 1 at pre-dose, 0.25, 0.5, 1, 1.083, 1.25, 1.5, 1.75,2, 3, 4, 6, 8, 12 hrs; Day 2 at 24 and 36 hrs; Day 3 at 48hrs.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage bioavailability
Arm/Group | Edaravone Oral Suspension
Number analyzed (Participants) | 42
percentage bioavailability | 57.3 (12.6)

20. Secondary Outcome: AUC0-t of Sulfate and Glucuronide Conjugates After Oral and Intravenous Administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
ng·h/mL
  Sulfate conjugate | 20031 (5255) | 15024 (3576)
  Glucuronide Conjugate | 3914 (730) | 2285 (481)

21. Secondary Outcome: AUC0-inf of Sulfate and Glucuronide Conjugates After Oral and Intravenous Administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
ng·h/mL
  Sulfate conjugate | 20055 (5256) | 15055 (3579)
  Glucuronide conjugate | 3924 (731) | 2295 (482)

22. Secondary Outcome: Cmax of Sulfate and Glucuronide Conjugates After Oral and Intravenous Administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
ng/mL
  Sulfate conjugate | 7291 (1898) | 4843 (817.8)
  Glucuronide conjugate | 2237 (388) | 1012 (235.7)

23. Secondary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions
Time Frame: Day 1 to 11
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
Number analyzed (Participants) | 42 | 42
Participants
  Number of Participants with Adverse events | 1 | 1
  Number of Participants with adverse drug reactions | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 11
Arm/Group | Edaravone Oral Suspension | Edaravone IV Formulation
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 1/42 | 1/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edaravone Oral Suspension (N=42) | Edaravone IV Formulation (N=42)
Constipation (Gastrointestinal disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT04493281/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT04493281/SAP_001.pdf